CLINICAL TRIAL: NCT06869473
Title: A Single-arm Phase II Study of Cetuximab Plus Platinum and Taxane-based Chemotherapy Followed by AVElumab and Cetuximab as First-line Therapy for Recurrent/Metastatic (R/M) Head and Neck Squamous Cell Carcinoma (HNSCC) Patients With PD-L1 Combined Positive Score (CPS)≥1≤19: the Immunotherapy Sequenc
Brief Title: Cetuximab Plus Platinum and Taxane-based Chemotherapy, Followed by Avelumab and Cetuximab, as First-line Treatment for Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma (HNSCC) Patients With a PD-L1 Combined Positive Score (CPS)≥1≤19.
Acronym: AVEC-119
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Collaborators: Merck Serono S.P.A., Italy (Industry); Clinical Research Technology S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVEC-119; 2024-512053-24-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-27; First posted 2025-03-11 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC); Recurrent Head and Neck Cancer; Metastatic Head and Neck Cancer
Keywords: Head and Neck Neoplasms; Squamous Cell Carcinoma; Cetuximab; Avelumab; Anti-EGFR Therapy; Platinum-Based Chemotherapy; Taxane-Based Chemotherapy; PD-L1 Combined Positive Score (CPS)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Cetuximab; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single-arm (Experimental): in-label induction therapy with three cycles of TPE (Paclitaxel, platinum-based compound, Cetuximab), followed, only in patients who are (partially or completely) responders and stable, by a maintenance therapy with the combination of AVEC (Avelumab, an anti-PD-L1 drug, plus Cetuximab, an anti-EGFR drug) extended until disease progression, unacceptable toxicity, or patient withdrawal.
  Interventions: Drug: Cetuximab/avelumab

INTERVENTIONS:
Drug: Cetuximab/avelumab — Study Maintenance therapy: AVEC (each cycle every 2 weeks) Cetuximab will be administered at 500 mg/m2 dose (as a 2-hour intravenous infusion) every 2 weeks until disease progression or unacceptable side effects.
  Cetuximab will be administered by IV infusion over 120 minutes. The initial dose should be given slowly and speed of infusion must not exceed 5 mg/min.
  Avelumab will be administered at 800 mg flat dose (as a 1-hour intravenous fusion) every 2 weeks until disease progression or unacceptable side effects.

SUMMARY:
This phase II interventional clinical trial aims to evaluate whether combining cetuximab and avelumab, after three cycles of platinum and taxane-based chemotherapy, can improve treatment outcomes for patients with recurrent or metastatic (R/M) head and neck squamous cell carcinoma (HNSCC) with a PD-L1 combined positive score (CPS) between 1 and 19. Specifically, the study seeks to determine if this approach can increase the 6-month progression-free survival (PFS) rate from 40% to 55%.

The trial will include adult patients with confirmed R/M HNSCC, who have not previously received systemic therapy for their advanced disease. By testing this sequential treatment strategy, researchers hope to improve outcomes for this specific patient population, which has shown poorer responses to existing immunotherapy options compared to those with higher PD-L1 expression levels.

Participants will first undergo an induction phase, consisting of three cycles of chemotherapy with paclitaxel, platinum (cisplatin or carboplatin), and cetuximab. After this initial treatment, they will move to a maintenance phase, where they will receive avelumab and cetuximab every two weeks until disease progression or the occurrence of unacceptable side effects.

The study aims to answer several key questions:

Can this treatment approach improve progression-free survival at 6 months? What impact does it have on overall survival, response rates, and the duration of response? Is this combination therapy safe and well-tolerated? In addition to the treatment itself, participants will be asked to provide blood and tumor tissue samples for translational research, helping scientists better understand how biomarkers influence treatment response. Regular follow-up assessments will also be conducted to monitor disease progression and overall health.

By testing this innovative treatment sequence, researchers hope to bridge the gap between different PD-L1 subgroups, potentially offering a more effective and personalized approach for patients with R/M HNSCC.

DETAILED DESCRIPTION:
This clinical study, titled AVEC-119, is a phase II, single-arm trial designed to evaluate the efficacy and safety of an innovative treatment approach for recurrent and metastatic head and neck squamous cell carcinoma (R/M HNSCC). The study aims to explore whether reversing the conventional immunotherapy sequence-initiating treatment with anti-EGFR-based chemotherapy induction followed by checkpoint inhibition-can significantly improve patient outcomes. The therapy consists of Cetuximab in combination with platinum- and taxane-based chemotherapy during the induction phase, followed by maintenance therapy with Avelumab (a PD-L1 inhibitor) and Cetuximab.

Objective:

The primary goal of this study is to determine whether this unique sequential treatment strategy can enhance six-month progression-free survival (PFS) rates in patients with PD-L1 CPS≥1≤19 R/M HNSCC. By leveraging the potential immune-stimulating effects of anti-EGFR therapy and chemotherapy, followed by immunotherapy maintenance, the study aims to improve overall survival and tumor response rates compared to standard treatment regimens.

Rationale:

Over the past decade, immune checkpoint inhibitors (ICIs) have reshaped the first-line treatment landscape for R/M HNSCC. Findings from the Keynote-048 trial demonstrated that pembrolizumab, administered alone or in combination with chemotherapy, led to prolonged overall survival (OS) compared to the EXTREME regimen (Cetuximab + platinum + 5-FU). However, these improvements were primarily observed in patients with a PD-L1 CPS≥20. In contrast, those with PD-L1 CPS between 1 and 19 did not achieve significant benefits in progression-free survival (PFS) or overall response rate (ORR), highlighting an area of unmet clinical need.

Previous studies have demonstrated that regimens incorporating Cetuximab with platinum- and taxane-based chemotherapy offer comparable efficacy and superior safety profiles compared to platinum + 5-FU regimens. Furthermore, taxanes and anti-EGFR therapies may enhance anti-tumor immune responses, priming the tumor microenvironment for subsequent immunotherapy.

AVEC-119 aims to harness this synergy by first reducing the tumor burden and modulating the immune microenvironment through induction therapy with Cetuximab and chemotherapy, followed by immune checkpoint inhibition with Avelumab in combination with Cetuximab. This innovative treatment approach is designed to improve response rates and extend survival in patients who typically derive limited benefit from standard checkpoint inhibitors.

Study Design:

Study Type: Multicenter, single-arm, phase II trial Participating Sites: 8 specialized oncology centers in Italy Target Population: Patients with R/M HNSCC and PD-L1 CPS between 1 and 19 Planned Enrollment: A total of 67 patients

Treatment Plan:

Induction Phase (TPE - 9 weeks):

* Paclitaxel: 175 mg/m² IV infusion every 21 days (3 cycles)
* Cisplatin: 75 mg/m² IV infusion every 21 days (3 cycles) (Carboplatin AUC 5 may be substituted for patients with renal impairment or neuropathy)
* Cetuximab: Initial dose of 400 mg/m² IV infusion, followed by 250 mg/m² weekly for 3 cycles

Maintenance Phase (AVEC - Until Disease Progression or Toxicity):

* Avelumab: 800 mg IV every 2 weeks
* Cetuximab: 500 mg/m² IV every 2 weeks Translational Research and Biomarker Analysis AVEC-119 integrates a comprehensive translational research component aimed at unraveling the molecular mechanisms underlying treatment response and resistance.

The study will:

* Conduct pre-treatment gene expression (GE) analysis in tumor samples to explore correlations between hypoxia, immune activity, and response to therapy.
* Utilize single-cell sequencing to track immune cell population changes in blood samples collected at four critical time points: pre-TPE, post-TPE, during maintenance (6 months), and at disease progression.
* Investigate whether the hypoxic and immune landscape of tumors shifts following EGFR inhibition, potentially enhancing response to subsequent PD-L1 blockade.

Ethical and Regulatory Aspects

* The study adheres to Good Clinical Practice (GCP) standards and has obtained approval from the relevant ethics committees.
* All participants provide informed consent prior to enrollment.
* Patient safety is continuously monitored, with predefined stopping criteria in place should unacceptable toxicity levels arise.

Conclusion AVEC-119 represents a paradigm shift in the treatment of R/M HNSCC, particularly for patients with PD-L1 CPS between 1 and 19, a group that has historically exhibited suboptimal responses to checkpoint inhibitors. By reversing the conventional immunotherapy sequence-priming the immune system with a chemotherapy/EGFR-targeted induction before introducing checkpoint blockade-this study aims to achieve higher response rates, prolong progression-free survival, and shed new light on tumor-immune dynamics. If successful, this approach may redefine first-line treatment strategies for a challenging subset of head and neck cancer patients, offering new hope and improved clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects able to sign the informed consent and ≥18 y-old.
2. Histologically or cytologically confirmed diagnosis of HNSCC.
3. Confirmed R/M HNSCC (i.e. oral cavity, oropharynx, larynx, hypopharynx) not suitable for curative loco-regional therapy.
4. PD-L1 CPS≥1≤19 (assessment allowed either on primary and/or recurrent/metastatic site of disease).
5. Measurable disease according to RECIST Criteria 1.1.6. Subjects should not have had prior systemic therapy administered in the R/M HNSCC setting.

7.Systemic therapy that was completed more than 6 months prior to signing consent, if given as a part of multimodal curative treatment for locally advanced disease, is allowed.

8.ECOG Performance Status (PS) 0-1. 9.Adequate bone marrow function: neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, hemoglobin ≥ 9 g/dL.

10.Adequate liver function: total bilirubin level < 1.5 X Upper Limit of Normal (ULN) (except for known medical reason not interfering with liver function, such as Gilbert syndrome), AP, GGT <3 x ULN and AST and ALT levels ≤ 2.5 × ULN.

11.Adequate renal function: calculated or analyzed creatinine clearance ≥ 30 mL/min.

12.Archival or fresh tissue of primary disease (i.e. T and/or N and/or M) OR recurrent/metastatic disease available at baseline (before starting TPE) (available as Formalin-Fixed Paraffin-Embedded - FFPE - or as unstained 10-20 slices).

13.Participants have to provide peripheral blood samples (at least 8-10 mL stored in EDTA) according the timing described in the translational part of the current protocol.

14.Palliative radiotherapy and/or surgery within 4 weeks before the study entry are allowed.

15.Symptomatic peripheral neuropathy NCI-CTC v5.0 grade ≥ 2 and / or ototoxicity grade ≥ 2, (except for cases in which ototoxicity is due to trauma or tumor-related mechanical impairment) or creatinine clearance < 60 mL/min are acceptable and they must be approached with carboplatin (instead of cisplatin) since the trial start.

Exclusion criteria:

1. Nasopharyngeal, salivary gland, nasal sinus, and non-melanoma skin cancers are not allowed.
2. Life expectancy lower than 3 months according to the judgement of trial investigator is not allowed.
3. Previous chemotherapy, or biological therapy (i.e. Cetuximab), or immunotherapy administered for R/M setting of HNSCC is not allowed.
4. Diagnosis of immunodeficiency or subjects receiving systemic steroid therapy (> 10 mg/day of prednisone or equivalent) or any other form of immunosuppressive therapy within 30 days prior to start of study treatment which cannot be interrupted.
5. Known allergic/hypersensitivity reaction to investigational products or any component in their formulations.
6. Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
7. Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with type I diabetes, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
8. Any diagnosed and/or treated additional malignancy within 5 years before the study entry with the exception of: curatively treated basal cell carcinoma of the skin, curatively treated squamous cell carcinoma of the skin, curatively treated prostate cancer, curatively resected in situ cervical cancer, and curatively resected in situ breast cancer.
9. Subjects with a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subjects' participation for the full duration of the trial, or is not in the best interest of the subject to participate, according to the opinion of the treating investigator.
10. Significant neurologic or known psychiatric or substance abuse disorders that would interfere with cooperation and the requirements of the trial.
11. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (≤6 months prior to enrollment), myocardial infarction (≤6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
12. Prior organ transplantation including allogenic stem-cell transplantation.
13. Active uncontrolled infection requiring systemic therapy (i.e. I.V. antibiotics).
14. Known history of testing positive for HIV or known acquired immunodeficiency syndrome.
15. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening tests positive).
16. Live vaccination within 30 days of planned start of study treatment (inactivated vaccines are allowed).
17. Pregnancy (absence of pregnancy must be confirmed by negative serum or urine pregnancy test - ß-HCG - for women of childbearing potential) and/or breast-feeding are not allowed. Subjects of childbearing potential willing to use effective contraceptive method [Pearl Index < 1; e.g. oral contraceptive (pill), hormone spiral, hormone implant, transdermal patch, a combination of two barrier methods (condom and diaphragm), sterilization, sexual abstinence] for the entire study duration and 30 days post-dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2027-08-20 (Estimated); Study Completion 2028-02-20 (Estimated)

PRIMARY OUTCOMES:
6-months (6m)-Progression Free Survival | 6-months from baseline
  The increase of the 6-months (6m)-Progression Free Survival intended as the time from baseline until first evidence of disease progression or death, from 40% to 55% in PD-L1 CPS≥1≤19 R/M HNSCC patients.

SECONDARY OUTCOMES:
overall survival (OS) | From date of enrollment until the date of first documented until the date of death from any cause, assessed up to 12 months from last subject in
  Overall Survival (OS) of TPE followed by avelumab and cetuximab in PD-L1 CPS≥1≤19 R/M HNSCC patients.
overall response rate (ORR) | Up to 12 months
  overall response rate (ORR) of cetuximab plus platinum and taxane-based chemotherapy followed by avelumab and cetuximab maintenance.
safety of cetuximab plus platinum and taxane-based chemotherapy | up to 12 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
duration of response (DOR) | Up to 12 months
  duration of response (DOR) of cetuximab plus platinum and taxane-based chemotherapy followed by avelumab and cetuximab maintenance.

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (8):
  - Ospedale Oncologico "A. Businco" ARNAS BROTSU, Cagliari, CAGLIARI
  - Azienda Ospedaliero-Universitaria Policlinico "G. Rodolico-S. Marco, Catania, CATANIA
  - Azienda Ospedaliero-Universitaria Careggi, Florence, FIRENZE
  - Fondazione IRCCS Istituto Nazionale dei Tumori (INT) di Milano, Milan, Milano
  - Irccs Humanitas Research Hospital, Rozzano, Milano
  - Irccs Fondazione G. Pascale, Napoli, Napoli
  - AOU Luigi Vanvitelli, Napoli, NAPOLI
  - Azienda Ospedaliero-Universitaria Sant'Andrea, Roma, roma

IPD SHARING:
Plan to Share IPD: No
due to technical issues